CLINICAL TRIAL: NCT02540837
Title: Analgesic Effect of an Obturator Nerve Block Combined With a Femoral Nerve Block Compared With Femoral Nerve Block Alone in Patients With Hip Fracture
Brief Title: Obturator and Femoral Nerve Block in Patients With Hip Fracture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol2_2tdn
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Experimental): Obturator nerve block
  Interventions: Drug: Bupivacaine
- Saline (Placebo Comparator): Saline is injected as a placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — Obturator nerve block
  Other Names: Active nerve block
  Arms: Bupivacaine
Drug: Saline — Obturator nerve block with saline(placebo)
  Other Names: Placebo
  Arms: Saline

SUMMARY:
A higher number than expected of patients with hip fracture have only insufficient analgesic effect of a femoral nerve block, which is the nerve block commonly used for this group of patients. One of the possible causes of this failure to provide analgesia from a single nerve block could be the that other nerves are involved in transmitting the pain signal. One of the nerves that is believed to give off branches to the hip is the obturator nerve.

With ultrasound it is possible to make a selective proximal nerve block of the obturator nerve.

The aim of this trial is to test the analgesic effect of a femoral nerve block i combination with an obturator nerve block compared to femoral nerve block alone in a randomized and placebo controlled design.

DETAILED DESCRIPTION:
A higher number than expected of all patients with hip fracture have only insufficient analgesic effect of a femoral nerve block. One of the possible causes of this failure to provide analgesia from a single nerve block could be the that other nerves are involved in transmitting the pain signal. One of the nerves that is believed to give off branches to the hip is the obturator nerve. Earlier it was believed that the so called '3-in-1-block' or the iliac fascia compartment block would anesthetize also the obturator nerve, and these two nerve blocks have been uses extensively in the emergency ward for preoperative analgesia. Today that is not believed to be true and consequently is the part of the obturator nerve in patients with hip fracture unknown.

With ultrasound it is possible to make a selective proximal nerve block of the obturator nerve before it branches into an anterior and a posterior branch. A selective nerve block of the obturator nerve to access its effect in patients with hip fracture has to our knowledge never been done.

The aim of this trial is to test the analgesic effect of a femoral nerve block i combination with an obturator nerve block compared to femoral nerve block alone in a randomized and placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of hip fracture
* Age ≥ 55 years
* Mentally capable of comprehending and using verbal pain score
* Mentally capable of differentiating between pain from the fractured hip and pain from other locations
* Mentally capable of understanding the given information
* Arrival in the emergency room at times when one of the doctors who do the nerve blocks for this investigation are on call
* Verbal numeric pain scale score (NRS 0-10) > 5 with a dynamic test OR NRS > 3 at rest
* Patients informed consent

Exclusion Criteria:

* Hip fracture not confirmed by x-ray
* Weight < 40 kg
* Patient has previously been included in this trial
* If the patient wishes to be excluded
* Allergy to local anesthetics or adrenocortical hormone
* Visible infection in the area of the point of needle injection

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Success rate of successful analgesia, measured with numeric rating scale(NRS) 0-10 with 0=no pain and 10=worst pain. Successful analgesia = NRS<4 at rest and NRS <6 with passive movement of the fractured leg. | 30 minutes
  Success rate of successful analgesia compared between the groups

SECONDARY OUTCOMES:
Median pain score (NRS 0-10) | 30 minutes
  Median pain score 30 minutes after the nerve blocks compared between the groups
Median change in pain score (NRS 0-10) | 30 minutes
  Median change in pain score 30 minutes after the nerve blocks compared between the groups
Course in pain reduction | 30 minutes
  Course in pain reduction during the 30 minutes after the nerve blocks
Time to sufficient analgesia | 30 minutes
  Time from ended injection until sufficient analgesia
Frequency of anesthesia in the skin area of the saphenous nerve | 30 minutes
  Frequency of anesthesia in the skin area innervated by the saphenous nerve
Frequency of anesthesia in the skin area of the anterior cutaneous branches of the femoral nerve | 30 minutes
  Frequency of anesthesia in the skin area of the anterior cutaneous branches of the femoral nerve
Localization of the worst pain before block | 0 minutes
  Localization of the worst pain before any nerve blocks
Localization of the worst pain after block | 30 minutes
  Localization of the worst pain 30 minutes after the nerve blocks
Discomfort during nerve block procedures (score 0-10, 0=no discomfort) | 5 minutes
  Discomfort during the nerve block procedures compared between procedures
Satisfaction (0-10, 0= very unsatisfactory) | 30 minutes
  Patient satisfaction with the pain treatment
Frequency of ultrasound visualization of femoral nerve | 5 minutes
  Frequency of patients with possible ultrasound visualization af the femoral nerve
Frequency of ultrasound visualization of obturator injection site | 5 minutes
  Frequency of patients with possible ultrasound visualization of the obturator nerve block injection site
Time spend on femoral nerve block | 5 minutes
  Time spend on conducting the femoral nerve block
Time spend on obturator nerve block | 5 minutes
  Time spend on conducting the obturator nerve block
Total morphine equivalent dose of opioid from the time of nerve block to operation | Approximately 24 hours in average
  Total morphine equivalent dose of opioid from the time of nerve block until the time of operation
Total morphine equivalent dose of opioid/time from the time of nerve block to operation | Approximately 24 hours in average
  Total morphine equivalent dose of opioid/time from the time of nerve block until the time of operation
Total morphine equivalent dose of opioid in the first 10 hours after nerve block | 10 hours
  Total morphine equivalent dose of opioid given in the first 10 hours after nerve block
Total morphine equivalent dose of opioid/time in the first 10 hours after nerve block | 10 hours
  Total morphine equivalent dose of opioid/time given in the first 10 hours after nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Bendtsen, Ph.d., Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark